CLINICAL TRIAL: NCT00171951
Title: Extension to a Multicenter, Open-label Study to Assess the Safety and Efficacy of 600 μg SOM230, Administered Subcutaneously, Bid in Patients With Cushing's Disease
Brief Title: Extension Study to Assess the Safety and Efficacy of Pasireotide in Participants With Cushing's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230B2208E1; 2004-002407-32 (EudraCT Number)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Cushing Disease
Keywords: Cushing's disease; ACTH; Cortisol; ACTH dependent Cushing's disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — pasireotide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC (Experimental): Participants received pasireotide 600 micrograms (μg) twice daily (BID) subcutaneously (SC) to achieve or maintain urinary free cortisol (UFC) normalization. If UFC levels were increased at any time, participants received 900 μg BID SC, until no safety or tolerability concerns were observed as per investigators assessment. If the participant was unable to tolerate the 900 μg BID, dosing of 600 μg three times a day was given.
  Interventions: Drug: Pasireotide

INTERVENTIONS:
Drug: Pasireotide — Pasireotide 600 μg or 900 μg was administered as an SC injection.
  Other Names: SOM230

SUMMARY:
Cushing's disease is a rare serious condition that is caused by an adrenocorticotropic hormone (ACTH) secreting pituitary adenoma. This study assessed the long-term safety and efficacy of pasireotide in participants with Cushing's disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have completed the 15 days of Pasireotide treatment in the CSOM230B2208 study and have achieved normalization of 24-hour urinary free cortisol. Participants who did not achieve normalization of 24 -hour urinary free cortisol may be enrolled if in the opinion of the investigator the participant is getting significant clinical benefits from treatment with Pasireotide .
* The participant did not experience any unacceptable adverse events of tolerability issues during the original 15 day treatment.
* Female participants of childbearing potential who have not undergone clinically documented total hysterectomy and/or ovariectomy or tubal ligation must agree to use barrier contraception throughout the course of the extension study, and for one month after the study has ended.

Exclusion Criteria:

* Participant who have developed poorly controlled diabetes mellitus as indicated by ketoacidosis or hemoglobin (Hgb) A1C (HgbA1C) > 10 since starting [study CSOM230B2208].
* Participant with persistent alanine aminotransferase (ALT)/ aspartate transaminase (AST) or alkaline phosphatase levels more than 2.5X upper limit of normal (ULN), serum creatinine > 2.0 X ULN, serum bilirubin > 2 X ULN.
* Participant with abnormal coagulation (Prothrombin time (PT) and partial thromboplastin time (PTT) elevated by 30% above normal limits), white blood cells (WBC) <3.0x1'000'000'000/L; Hgb <12.0g/dL for females, Hgb <13.0g/dL for males; PLT <100x1'000'000'000/L.

Other protocol-defined inclusion / exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-08-13 (Actual); Primary Completion 2013-07-08 (Actual); Study Completion 2013-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticlas, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Oregon Health & Sciences University Dept.ofOregonHealth&SciencesU., Portland, Oregon
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
- Novartis Investigative Site, Paris, France
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, München
- Novartis Investigative Site, Ancona, AN, Italy
- Novartis Investigative Site, Belfast, United Kingdom

REFERENCES:
- [Result] Boscaro M, Bertherat J, Findling J, Fleseriu M, Atkinson AB, Petersenn S, Schopohl J, Snyder P, Hughes G, Trovato A, Hu K, Maldonado M, Biller BM. Extended treatment of Cushing's disease with pasireotide: results from a 2-year, Phase II study. Pituitary. 2014 Aug;17(4):320-6. doi: 10.1007/s11102-013-0503-3. PMID 23943009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included participants with Cushing's disease who received 15 days of pasireotide treatment in the Core Study CSOM230B2208 (NCT00088608). This study was an extension study of the Core Study.
Period: Overall Study
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Started | 19
Completed | 3
Not Completed | 16
Not completed — Adverse Event | 1
Not completed — Abnormal Laboratory Values | 2
Not completed — Unsatisfactory Therapeutic Effect | 3
Not completed — Participants Withdrew Consent | 3
Not completed — New Cancer Therapy | 5
Not completed — Reason not Specified | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who completed 15 days of treatment in Core study and experienced significant clinical benefit from treatment and received at least 1 dose in the Extension Period.
Groups:
- Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC: Participants received pasireotide 600 μg BID SC to achieve or maintain UFC normalization. If UFC levels were increased at any time, participants received 900 μg BID SC, until no safety or tolerability concerns were observed as per investigators assessment. If the participant was unable to tolerate the 900 μg BID, dosing of 600 μg three times a day was given.
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders With Mean Urinary Free Cortisol (UFC) Within Normal Limits
Description: A participant was considered a responder if the mean UFC from the two 24-hour urine samples collected at Month 6 was within normal limits. The normal range for UFC is 55 to 276 nmol/day.
Time Frame: Month 6
Population: Primary Efficacy Population included participants from ITT whose mean UFC at core-baseline, based on at least 2 UFC samples, was >1.0x upper limit of normal (ULN) or for whom the one and only UFC sample available at baseline was >2.0xULN.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 18
percentage of responders | 22.2 [6.4 to 47.6]

2. Primary Outcome: Change From Baseline in Mean Urinary Free Cortisol (UFC)
Description: 24-hour urine samples were collected to obtain mean UFC measurements. A negative mean change from baseline indicates improvement.
Time Frame: Core Baseline, Days 14/15 (Core study), Months 6, 12, 24 and 102
Population: Primary Efficacy Population included participants from ITT whose mean UFC at core-baseline, based on at least 2 UFC samples, was >1.0x ULN or for whom the one and only UFC sample available at baseline was >2.0xULN. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: nanomoles per 24 hours (nmol/24h)
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 18
nanomoles per 24 hours (nmol/24h)
  Core Baseline: number analyzed (Participants) | 17
  Core Baseline | 1219.74 (752.9)
  Change from Core Baseline to Day 14/Day 15: number analyzed (Participants) | 16
  Change from Core Baseline to Day 14/Day 15 | -710.57 (740.6)
  Change from Core Baseline to Month 6: number analyzed (Participants) | 10
  Change from Core Baseline to Month 6 | -801.85 (819.4)
  Change from Core Baseline to Month 12: number analyzed (Participants) | 4
  Change from Core Baseline to Month 12 | -1202.1 (1084.1)
  Change from Core Baseline to Month 24: number analyzed (Participants) | 4
  Change from Core Baseline to Month 24 | -1241.1 (925.6)
  Change from Core Baseline to Month 102: number analyzed (Participants) | 1
  Change from Core Baseline to Month 102 | -2417.0 (NA) — Due to one participant available for analysis standard deviation (SD) was not estimable.

3. Secondary Outcome: Number of Participants Who Had At Least One Adverse Event (AE)
Description: An AE was any undesirable sign, symptom or medical condition occurring after starting study drug even if the event is not considered to be related to study drug. AEs were assessed according to incident dose group: Pasireotide 1200 μg sc total daily dose (TDD), Pasireotide 1800 μg SC TDD and Pasireotide SC Any Dose. The incident dose for an AE was the last total daily dose administered on or prior to the AE onset date.
Time Frame: Up to approximately 106 months
Population: Safety Population included participants from ITT Population. ITT Population included participants who completed 15 days of treatment in the Core study, experienced significant clinical benefit without any unacceptable AEs, and received at least 1 dose in the extension period.
Measure: Count of Participants; unit: Participants
Groups:
- Pasireotide 600 μg BID SC: Participants received pasireotide 600 μg BID SC, to achieve or maintain UFC normalization.
- Pasireotide 900 μg BID SC: Participants received 900 μg BID SC if UFC levels were increased at any time, until no safety or tolerability concerns were observed as per investigators assessment. If the participant was unable to tolerate the 900 μg BID, dosing of 600 μg three times a day was given.
Arm/Group | Pasireotide 600 μg BID SC | Pasireotide 900 μg BID SC
Number analyzed (Participants) | 19 | 8
Participants | 19 | 8

4. Secondary Outcome: Change From Baseline in Serum Cortisol Levels
Description: Blood samples were withdrawn to obtain the serum cortisol levels. A negative change from baseline indicates improvement.
Time Frame: Core Baseline, Day 15 (Core study), Months 6, 12, 24, and Month 105 (end of the study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanomoles per liters (nmol/L)
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 18
nanomoles per liters (nmol/L)
  Core Baseline | 723.60 (221.5)
  Change from Core Baseline to Day 15 | -25.96 (125.1)
  Change from Core Baseline to Month 6: number analyzed (Participants) | 11
  Change from Core Baseline to Month 6 | -150.60 (308.9)
  Change from Core Baseline to Month 12: number analyzed (Participants) | 5
  Change from Core Baseline to Month 12 | -66.06 (301.9)
  Change from Core Baseline to Month 24: number analyzed (Participants) | 4
  Change from Core Baseline to Month 24 | -227.53 (283.1)
  Change from Core Baseline to Month 105: number analyzed (Participants) | 1
  Change from Core Baseline to Month 105 | -166.00 (NA) — Due to one participant available for analysis SD was not estimable.

5. Secondary Outcome: Plasma Trough Concentrations (Ctrough) of Pasireotide in UFC Responders
Description: Participants with Cushing's disease were considered responders if mean UFC levels from the 24-hour urine collections at Day 15 (Core study) and at extension Month 6, were within normal limits. Ctrough levels of pasireotide were measured at Day 15 of Core study and Month 6.
Time Frame: Day 15 (Core study) and Month 6
Population: Pharmacokinetic (PK) Population included participants from ITT who had at least one post dosing PK assessment up to the implementation of Amendment 2 when no further blood samples were collected for PK assessment (24 May 2007).
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 4
nanograms per milliliter (ng/mL)
  Day 15 (Core Study) | 7.0 (4.3)
  Month 6 | 17.4 (11.6)

6. Secondary Outcome: Change From Baseline in Plasma Adrenocorticotropic Hormone (ACTH) Levels
Description: Blood samples were withdrawn to obtain the ACTH levels. A negative change from baseline indicates improvement.
Time Frame: Core Baseline, Day 15 (Core study), Months 6, 12, 24 and Month 105 (end of the study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picomoles per litre (pmol/L)
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 18
picomoles per litre (pmol/L)
  Core Baseline | 13.72 (11.0)
  Change from Core Baseline to Day 15 | -1.28 (7.1)
  Change from Core Baseline to Month 6: number analyzed (Participants) | 11
  Change from Core Baseline to Month 6 | -3.36 (9.4)
  Change from Core Baseline to Month 12: number analyzed (Participants) | 5
  Change from Core Baseline to Month 12 | -3.60 (15.2)
  Change from Core Baseline to Month 24: number analyzed (Participants) | 4
  Change from Core Baseline to Month 24 | -4.50 (8.3)
  Change from Core Baseline to Month 105: number analyzed (Participants) | 1
  Change from Core Baseline to Month 105 | 0.00 (NA) — Due to one participant available for analysis SD was not estimable.

7. Secondary Outcome: Change From Baseline in Gene-expression and Protein in Blood and Urine for Biomarker Development
Time Frame: Baseline to end of the study
Population: We have exhausted all efforts to locate this data and it has since been destroyed, therefore no data is available to report for this outcome measure.
Arm/Group | Pasireotide 600 μg BID SC or Ramp up Dose 900 μg BID SC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 106 months
Description: Safety Population included participants from ITT Population. ITT Population included participants who completed 15 days of treatment in the Core study, experienced significant clinical benefit without any unacceptable AEs, and received at least 1 dose in the extension period.
Arm/Group | Pasireotide 600 μg BID SC | Pasireotide 900 μg BID SC
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/19 | 2/8
Other Adverse Events (participants affected / at risk) | 19/19 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 600 μg BID SC (N=19) | Pasireotide 900 μg BID SC (N=8)
Urinary tract infection (Infections and infestations) | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide 600 μg BID SC (N=19) | Pasireotide 900 μg BID SC (N=8)
Diarrhoea (Gastrointestinal disorders) | 12 | 2
Nausea (Gastrointestinal disorders) | 12 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 3
Abdominal pain (Gastrointestinal disorders) | 8 | 2
Headache (Nervous system disorders) | 7 | 0
Injection site pain (General disorders) | 6 | 0
Asthenia (General disorders) | 4 | 1
Dizziness (Nervous system disorders) | 4 | 1
Fatigue (General disorders) | 5 | 0
Injection site pruritus (General disorders) | 5 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 4 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Hypertension (Vascular disorders) | 2 | 2
Hypotension (Vascular disorders) | 4 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1
Oedema peripheral (General disorders) | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Amenorrhoea (Reproductive system and breast disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Fungal skin infection (Infections and infestations) | 2 | 0
Glycosylated haemoglobin increased (Investigations) | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 0
Influenza (Infections and infestations) | 1 | 1
Influenza like illness (General disorders) | 2 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0
Injection site erythema (General disorders) | 2 | 0
Injection site oedema (General disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Oedema (General disorders) | 2 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood cortisol increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
Blood sodium increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1
Bone marrow oedema (Blood and lymphatic system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac murmur (Investigations) | 1 | 0
Chills (General disorders) | 1 | 0
Cyst (General disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Homocystinaemia (Congenital, familial and genetic disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypogonadism (Endocrine disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retinopathy hypertensive (Eye disorders) | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0
Tongue disorder (Gastrointestinal disorders) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Vulvovaginitis (Infections and infestations) | 1 | 0
Weight decreased (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.